CLINICAL TRIAL: NCT06614465
Title: Effect of a Multimodal Rehabilitation Programme on Epigenetic Biomarkers, Quality of Life, Sexual Function and Muscle Strength in Women With Dyspareunia and Endometriosis: Protocol for a Randomised Controlled Trial.
Brief Title: Multimodal Rehabilitation Programme on Epigenetic Biomarkers, Quality of Life, Sexual Function and Muscle Strength in Women With Dyspareunia and Endometriosis.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clínica INEBIR (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Endometriosis and dyspareunia
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Multidisciplinary Communication
Keywords: Endometriosis; Dyspareunia; Multimodal Rehabilitation; Epigenetic Biomarkers; Quality of life; Sexual Function; Muscle Strength
MeSH Terms: conditions — Endometriosis; Dyspareunia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1.Experimental Group (Experimental): The intervention group will receive a multimodal rehabilitation programme including therapeutic exercise, health education and manual therapy.
  Interventions: Other: Multimodal Rehabilitation
- 2.Control Group (No Intervention): The control group will not receive this intervention.

INTERVENTIONS:
Other: Multimodal Rehabilitation — The intervention will consist of 4 sessions of education in pain neuroscience, 4 sessions of therapeutic exercise and 4 sessions of manual therapy in the abdominopelvic area.
  Arms: 1.Experimental Group

SUMMARY:
This study aims to evaluate the impact of a multimodal rehabilitation programme on epigenetic biomarkers in blood, quality of life, sexual function and pelvic floor muscle strength and endurance in women with dyspareunia and endometriosis.

DETAILED DESCRIPTION:
Introduction: Endometriosis is a benign gynaecological disease that affects approximately 10% of women of childbearing age, causing chronic pelvic pain and profound dyspareunia, which significantly impairs quality of life. This study aims to evaluate the impact of a multimodal rehabilitation programme on epigenetic biomarkers, quality of life, sexual function and muscle strength in women with dyspareunia and endometriosis.

Study Design: Pilot of Randomised controlled clinical trial according to CONSORT and TIDieR guidelines. The study will run from January 2025 to January 2026.

Inclusion criteria: Women between 18 and 55 years old, diagnosed with endometriosis with dyspareunia and chronic pelvic pain, with the ability to communicate in Spanish, and approval of their gynaecologist.

Exclusion criteria: Neurological, oncological, autoimmune or serious psychiatric diseases that prevent exercise or manual therapy.

Sample Size: 20 women diagnosed with dyspareunia and endometriosis, randomly divided into two groups: 10 in the intervention group and 10 in the control group.

Intervention: The intervention group will receive a multimodal rehabilitation programme including therapeutic exercise, health education and manual therapy. The control group will not receive this intervention.

Primary results: Measurements will be taken at four key points in time: baseline (T0), 2 months (T1), 6 months (T2) and 12 months (T3). To assess the effect of the intervention on miR-21 levels in saliva, quality of life (SF-36 questionnaire), sexual function (FSFI), pain, and pelvic floor muscle strength (measured with Oxford and Perfect scales).

Second Results: Measurement of systemic inflammation by CRP and IL-6, hormone levels (oestrogen and progesterone), stress and psychological well-being (HADS), muscle strength (EPI-NO), adherence to treatment and satisfaction with the intervention.

Ethics and Privacy: The study will have the approval of the Ethics Committee of the University of Pablo de Olavide, following the Declaration of Helsinki and Spanish regulations (Law 14/2007 on Biomedical Research). Participants will sign an informed consent form, and the data will be managed in accordance with the Spanish Data Protection Act (Law 3/2018).

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with endometriosis
* Women with dyspareunia and chronic pelvic pain
* Ability to communicate fluently verbally and in writing in the language of the research team, in this case Spanish.
* Approval to participate in the study by your regular gynaecologist who is part of your diagnosis and treatment.

Exclusion Criteria:

* A neurological, oncological or autoimmune disease that prevents the participant from performing exercise.
* Any type of pathology that prevents the participant from performing exercise.
* A diagnosis of severe psychiatric or neurological disorders that do not allow the participant to follow orders.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
miR-21 | 1 month
  miR-21 levels in saliva
Quality of life | 1 month
  will be measured with the The Short Form-36 Health Survey (SF-36). A higher score indicates better health status.
Sexual Function | 1 month
  Will be measured with the Female Sexual Function Index (FSFI) questionnaire. A higher score indicates better sexual function.
Pelvic Floor Muscle Strength | 1 month
  Will be measured with Oxford and Perfect scale. A higher score indicates better Muscle Strength status.
Pain | 1 month
  Will be measured with Brief Pain Inventory (BPI) Questionnaire. A higher score indicates worse health status.

SECONDARY OUTCOMES:
Systemic inflammation | 1 month
  Will be measured with polymerase chain reaction (PCR).
Hormone Levels | 1 month
  Will be measured with blood test.
Psychological condition | 1 month
  Will be measured with Hospital Anxiety and Depression Scale (HADS). A higher score indicates worse health status.
satisfaction with the intervention | 1 month
  Will be measured with MedRisk questionnaire. The MedRisk Instrument for Measuring Patient Satisfaction With Physical Therapy Care. A higher score indicates greater disability or more pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Pablo de Olavide, Seville, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No